CLINICAL TRIAL: NCT03905590
Title: To Evaluate the Efficacy of Guided Tissue Regeneration in the Healing of Periapical Defects With Periodontal Communication :A Randomized Controlled Trial With 3D Analysis Using CBCT."
Brief Title: Efficacy of Guided Tissue Regeneration in the Healing of Periapical Defects With Periodontal Communication Using CBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RITIKA YADAV
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Apico Marginal Defects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periapical surgery with amniotic membrane (Experimental): periapical surgery will be done and amniotic membrane will be placed over the defect before closure of flap
  Interventions: Procedure: Periapical surgery with amniotic membrane
- periapical surgery without amniotic membrane (Active Comparator): periapical surgery will be done without the placement of amniotic membrane over the defect before closure of flap
  Interventions: Procedure: periapical surgery without amniotic membrane

INTERVENTIONS:
Procedure: Periapical surgery with amniotic membrane — periapical surgery will be done followed by amniotic membrane placement over the defect
  Arms: periapical surgery with amniotic membrane
Procedure: periapical surgery without amniotic membrane — periapical surgery will be done without placement of membrane over the defect.
  Arms: periapical surgery without amniotic membrane

SUMMARY:
Healing of the Apicomarginal defects will be checked by comparing 2 groups . In first group amniotic membrane will be applied over the defect before flap closure during surgery and in second group no GTR material will be applied. Healing of the lesions will also be compared 2 dimensionaly and 3 dimensionaly using CBCT

DETAILED DESCRIPTION:
Study Title: - To evaluate the efficacy of guided tissue regeneration in the healing of periapical defects with periodontal communication: A randomized controlled trial with 3D analysis using CBCT.

Rationale: - Healing of lesions with apicomarginal defects is often less satisfactory. Various studies and case reports have reported high success rate with the use of guided tissue regeneration technique. Only few clinical trials have evaluated the effect of guided tissue regeneration on the healing of apicomarginal defects. To best of our knowledge only two studies have conducted randomized controlled trial. However, no study has used CBCT for the assessment of healing in such type of lesions. So, this is the first randomized controlled trial studying the effect of guided tissue regeneration in the healing of periapical defects with periodontal communication using 3D radiological evaluation using CBCT.

Aim & Objectives: - 1. To evaluate the difference in the healing outcome of periapical defects with periodontal communication with or without the use of guided tissue regeneration technique 2. To evaluate the difference in the healing outcome derived from the assessment of 2D periapical radiographs and 3 D CBCT imaging.

Setting: - Study will be conducted in Post Graduate Institute of Dental Sciences, Rohtak in the department of Conservative Dentistry & Endodontics.

Study Design: - A randomized controlled trial Time Frame: - 12 to 18 months Population / Participants: - Patients of age 16 years (male/female) and above will be enrolled in the study.

Inclusion criteria: - Patients of age 16 years and above, Patients with no general medical contraindications for oral surgical procedures (ASA-I and ASA-II according to the classification of the American Society of Anesthesiologist's, periapical defect with periodontal communication, periodontal pocket >6mm with apicomarginal communication confined to buccal aspect of interproximal space or mid buccal aspect of the root ., -ve response to vitality test, failed previous root canal treatment with purulent discharge or failed previous surgery or recurrent episode of purulent discharge.

Exclusion criteria: -Presence of buccal bone on flap elevation, Unrestorable tooth, fractured /perforated roots, smokers, pregnant females and lactating mothers.

Sample size: - 30 patients (15 patients in each group) Methods: - Diagnosis of the lesion will be made clinically and radiographically, vitality will be checked by EPT, preoperative clinical evaluation will include, clinical attachment level, gingival marginal position and pocket depth. Marginal bone loss, width of bony crypt, height of the bony crypt, depth of the crypt and height of the buccal bone plate (if present) will be measured radiographically and at the time of surgery. Surgical procedures will be carried out under operating microscope with 8 × 16 magnification by the standardized treatment methods.

Outcome measures: - Follow up of patients will be carried out at 3, 6, 9 & 12 months and outcome measures will be assessed clinically by absence of signs and symptoms and 2 dimensionally using radiographs by Rud and Molven criteria for periapical healing and 3 dimensionaly using CBCT by modified PENN criteria at 12 months follow up for periapical healing and buccal bone level.

Statistical method: - The data will be entered into Microsoft Excel and analysed using SPSS (Statistical Package for Social Science) package for relevant statistical comparison. Distribution of data into normal and non-normal will be done by Kolmogorov-Smir-Nov test. If the data will be normal then student T test and paired T test will be applied for unpaired and paired data respectively. For categorical data Chi - square test will be applied. The interobserver analysis will be done by cohen kappa analysis.

If the data will be non-normal then Mann - Whitney and Wilcoxon rank sum test will be applied for unpaired and paired data respectively. For categorical data Chi - square test will be applied. The interobserver analysis will be done by cohen kappa analysis.

ELIGIBILITY:
Inclusion Criteria

1. Patients of age 16 years and above.
2. Patients with no general medical contraindications for oral surgical procedures (ASA-I and ASA-II according to the classification of the American Society of Anesthesiologist's.
3. periapical defect with periodontal communication.
4. Periodontal pocket >6mm with apicomarginal communication confined to buccal aspect of interproximal space or mid buccal aspect of the root.
5. Negative response to vitality test.
6. failed previous root canal treatment with purulent discharge or failed previous surgery or recurrent episode of purulent discharge.

Exclusion criteria: -

1. Presence of buccal bone on flap elevation.
2. Unrestorable tooth.
3. fractured /perforated roots.
4. smokers.
5. pregnant females and lactating mothers

   .

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
healing of periapical defects with periodontal communication with or without the use of guided tissue regeneration technique | BASE LINE TO 1YEAR
  Follow up of patients will be carried out at 3, 6, 9 & 12 months and outcome measures will be assessed clinically by absence of signs and symptoms and 2 dimensionally using radiographs by Rud and Molven criteria for periapical healing and 3 dimensionaly using CBCT by modified PENN criteria at 12 months follow up for periapical healing and buccal bone level.

SECONDARY OUTCOMES:
the difference in the healing outcome as observed derived from the assessment of 2D periapical radiographs and 3 D CBCT imaging. | BASE LINE TO 1 YEAR
  The comparison of healing will be done 2 dimensionaly and 3 dimensionaly

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India